CLINICAL TRIAL: NCT01861990
Title: Valproic Acid for Children With Recurrent and Progressive Brain Tumors
Brief Title: Valproic Acid in Childhood Progressive Brain Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Feasibility of the trial was proven to be absent.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Amy-Lee Bredlau, Director, Pediatric Brain Tumor Program, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA2013; IRG-97-219-14 (Other Grant/Funding Number: American Cancer Society Institutional Research Grant)
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Pediatric Brain Tumor; Glioma; Anaplastic Astrocytoma; Medulloblastoma; Glioblastoma
Keywords: Glioma; Glioblastoma; Pediatric; Child; Brain tumor; Astrocytoma; Medulloblastoma; PNET
MeSH Terms: conditions — Glioma; Astrocytoma; Medulloblastoma; Glioblastoma; Brain Neoplasms; Neuroectodermal Tumors, Primitive | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): All participants will be enrolled on to one, open-label arm. Participants will be treated with valproic acid in addition to standard of care therapy.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — All participants enrolled on valproic acid arm.
  Other Names: Valproate, VPA, Depakote, Depakote ER, Depakene

SUMMARY:
The study investigates valproic acid added to radiation and temozolomide therapy (standard of care) for progressive or recurrent pediatric brain tumors.

DETAILED DESCRIPTION:
Patients with progressive or recurrent pediatric brain tumors are administered valproic acid, an HDAC inhibitor, along with standard of care therapy (radiation and temozolomide) for induction therapy. Thereafter, patients will be able to continue on valproic acid and temozolomide therapy as long as the combination is well tolerated and the tumor is not progressing.

ELIGIBILITY:
Inclusion Criteria:

* Subject, parent, or guardian willing and able to give informed consent
* Recurrent or progressive pediatric brain tumor, with MRI evidence of disease
* Age at first diagnosis of brain tumor 1-21 years old
* Lansky or Karnofsky performance score of at least 50 at diagnosis

Exclusion Criteria:

* Pregnancy
* Prior intolerance to valproic acid
* History of use of temozolomide
* Use of enzyme inducing anticonvulsant medications (see appendix B)
* Known urea cycle disorder (e.g. ornithine transcarbamylase deficiency)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Completion of protocol | 2 months
  Number of participants completing the protocol will be measured.

SECONDARY OUTCOMES:
Time to progression | 2 months
  Participants will be evaluated for progression every 2 months while on the study.

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Bredlau, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Van Nifterik KA, Van den Berg J, Slotman BJ, Lafleur MV, Sminia P, Stalpers LJ. Valproic acid sensitizes human glioma cells for temozolomide and gamma-radiation. J Neurooncol. 2012 Mar;107(1):61-7. doi: 10.1007/s11060-011-0725-z. Epub 2011 Oct 26. PMID 22037799
- [Background] Asklund T, Kvarnbrink S, Holmlund C, Wibom C, Bergenheim T, Henriksson R, Hedman H. Synergistic killing of glioblastoma stem-like cells by bortezomib and HDAC inhibitors. Anticancer Res. 2012 Jul;32(7):2407-13. PMID 22753697
- [Background] Fu J, Shao CJ, Chen FR, Ng HK, Chen ZP. Autophagy induced by valproic acid is associated with oxidative stress in glioma cell lines. Neuro Oncol. 2010 Apr;12(4):328-40. doi: 10.1093/neuonc/nop005. Epub 2009 Oct 15. PMID 20308311
- [Background] Weller M, Gorlia T, Cairncross JG, van den Bent MJ, Mason W, Belanger K, Brandes AA, Bogdahn U, Macdonald DR, Forsyth P, Rossetti AO, Lacombe D, Mirimanoff RO, Vecht CJ, Stupp R. Prolonged survival with valproic acid use in the EORTC/NCIC temozolomide trial for glioblastoma. Neurology. 2011 Sep 20;77(12):1156-64. doi: 10.1212/WNL.0b013e31822f02e1. Epub 2011 Aug 31. PMID 21880994
- [Background] Masoudi A, Elopre M, Amini E, Nagel ME, Ater JL, Gopalakrishnan V, Wolff JE. Influence of valproic acid on outcome of high-grade gliomas in children. Anticancer Res. 2008 Jul-Aug;28(4C):2437-42. PMID 18751431